CLINICAL TRIAL: NCT07185633
Title: A Prospective, Single-Arm, Phase II Clinical Study of Gecacitinib-Corticosteroids as First-Line Treatment for Grade II-IV Acute Graft-Versus-Host Disease After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Study of Gecacitinib-corticosteroid as First-line Therapy for Grade II-IV Acute Graft Versus Host Disease
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bin Gu (Other)
Responsible Party: Sponsor-Investigator, Bin Gu, Associate Chief Physician, The First Affiliated Hospital of Soochow University
Organization: The First Affiliated Hospital of Soochow University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20250824101854977
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: aGVHD
Keywords: GVHD; JAKi
MeSH Terms: interventions — Methylprednisolone Hemisuccinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Gecacitinib-Corticosteroid as first-line therapy(Gecacitinib po. 50mg bid and Corticosteroid iv. 2mg/kg/d )
  Interventions: Drug: Gecacitinib-Corticosteroid; Drug: Methylprednisolone sodium succinate

INTERVENTIONS:
Drug: Gecacitinib-Corticosteroid — Gecacitinib po. 50mg bid at least 28 days
Drug: Methylprednisolone sodium succinate — Methylprednisolone sodium succinate IV 2mg/kg/d.

SUMMARY:
This trial employs a single-arm, single-center design, planning to enroll 25 patients diagnosed with grade II-IV aGVHD at one center. Patients meeting all inclusion criteria and no exclusion criteria will be enrolled. After enrollment, all patients will receive Gecacitinib combined with methylprednisolone sodium succinate for at least 28 days.

After 28 days of Gecacitinib treatment, patients evaluated by the investigator as achieving Complete Response (CR) or Partial Response (PR) may continue study treatment for up to 24 weeks. If patients experience intolerance, disease progression, or require new systemic therapy, treatment will be adjusted.

DETAILED DESCRIPTION:
All patients will receive the combined treatment of Gecacitinib and methylprednisolone sodium succinate in addition to the existing treatment regimen (Cyclosporin A 150~250 μg/L and/or Tacrolimus 5~12 μg/L) or other adjuvant treatments.

Dosage: Gecacitinib PO 50mg Bid; Methylprednisolone sodium succinate IV 2mg/kg/d.

After completing treatment, the Gecacitinib dose may be gradually reduced until discontinuation, per the investigator's discretion.The researchers adjusted the dosage of glucocorticoids according to the patient's condition: Methylprednisolone sodium succinate was gradually reduced.

If disease progresses (aGVHD grade increases by one level) during Gecacitinib treatment, the investigator should initiate other salvage therapy as clinically needed. If aGVHD efficacy evaluation does not reach Complete Response(CR) or Partial Response(PR) after 28 days of Gecacitinib, the investigator should initiate other systemic therapy as clinically needed.

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntarily sign informed consent form (ICF); age ≥18 years at ICF signing.
* 2. Recipients who underwent non-myeloablative, myeloablative, or reduced-intensity allo-HSCT using bone marrow or peripheral blood stem cells.
* 3. Have received systemic corticosteroid therapy for no more than 2 days (48 hours).
* 4. Documented myeloid and platelet engraftment: Absolute Neutrophil Count (ANC) >0.5 × 10⁹/L for 3 consecutive days, platelet count >20 × 10⁹/L for 7 consecutive days without transfusion support (use of growth factors, transfusion support allowed).
* 5. Clinical diagnosis of Grade II-IV aGVHD according to the MAGIC (Mount Sinai Acute GVHD International Consortium) criteria.
* 6. ECOG performance status 0-2.
* 7. Life expectancy greater than 4 weeks.
* 8. Able to swallow tablets.
* 9. Capable of complying with study and follow-up procedures.

Exclusion Criteria:

* 1. Having undergone ≥2 allo-HSCT procedures.
* 2. SR-aGVHD occurring after unplanned donor lymphocyte infusion (DLI) used for prophylactic treatment of malignancy relapse. *Note: Patients receiving planned DLI as part of the transplant procedure, not intended for managing malignancy relapse, may be included.*
* 3. Concurrent treatment with other JAK inhibitors.
* 4. Presence of active bleeding.
* 5. Diagnosed or suspected chronic GVHD.
* 6. Presence of uncontrolled active infection. Uncontrolled active infection is defined as: hemodynamic instability due to sepsis, or worsening of symptoms, signs, or radiographic findings due to infection. Persistent fever without symptoms or with stable symptoms is not considered an uncontrolled active infection.
* 7. Presence of unresolved toxicity or complications due to allo-HSCT (excluding aGVHD).
* 8. Any significant clinical or laboratory abnormality that may affect safety evaluation, such as:

  1. Uncontrolled diabetes (fasting blood glucose >13.9 mmol/L);
  2. Hypertension that cannot be controlled to within SBP <160 mmHg and DBP <100 mmHg with two or more antihypertensive agents;
  3. Peripheral neuropathy (NCI-CTCAE v5.0 Grade 2 or higher).
* 9. History of NYHA Class III or IV congestive heart failure, uncontrolled or unstable angina, myocardial infarction, cerebrovascular accident, or pulmonary embolism within 6 months before screening.
* 10. Arrhythmia requiring treatment at screening, or QTc interval (QTcB) >480 ms.
* 11. Significant renal impairment at screening (serum creatinine >1.5 × ULN).
* 12. Pre-transplant diagnosed gastrointestinal ulcers, history of gastric/intestinal resection surgery, or other conditions potentially affecting drug absorption.
* 13. Surgery within 4 weeks before screening without full recovery.
* 14. Cholestatic disease or hepatic sinusoidal obstruction syndrome/veno-occlusive disease (SOS/VOD) at screening (defined as persistent bilirubin abnormality and progressive organ dysfunction not due to GVHD).
* 15. Active uncontrolled viral infection at screening, e.g., CMV, EBV, HIV (anti-HIV antibody positive), HBV (HBsAg positive, HBV-DNA positive), HCV (anti-HCV antibody or HCV-RNA positive).
* 16. History of active tuberculosis within 6 months before screening.
* 17. Epilepsy or use of psychotropic/sedative drugs at screening.
* 18. Women planning pregnancy, pregnant, or breastfeeding, or patients unable to use effective contraception throughout the trial; male patients unwilling to use condoms during treatment and for 2 days (approx. 5 half-lives) after the last dose.
* 19. History of other malignancies within the past 5 years, excluding the malignancy for which transplant was performed.
* 20. Other severe comorbidities deemed by the investigator to potentially affect patient safety or compliance.
* 21. Suspected allergy to gecacitinib, drugs of the same class, or any excipients.
* 22. Participation in other investigational drug or medical device clinical trials within 4 weeks before screening.
* 23. Any other condition considered by the investigator to preclude participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) for aGVHD at Day 28 of treatment | Day 28
  Defined as the percentage of patients achieving Complete Response (CR) + Partial Response (PR) at Day 28

REFERENCES:
- [Result] Dou L, Zhao Y, Yang J, Deng L, Wang N, Zhang X, Liu Q, Yang Y, Wei Z, Wang F, Jiao Y, Li F, Luan S, Hu L, Gao S, Liu C, Liu X, Yan J, Zhang X, Zhou F, Lu P, Liu D. Ruxolitinib plus steroids for acute graft versus host disease: a multicenter, randomized, phase 3 trial. Signal Transduct Target Ther. 2024 Oct 23;9(1):288. doi: 10.1038/s41392-024-01987-x. PMID 39438467
- [Result] Dou L, Peng B, Li X, Wang L, Jia M, Xu L, Li F, Liu D. Ruxolitinib-corticosteroid as first-line therapy for newly diagnosed high-risk acute graft versus host disease: study protocol for a multicenter, randomized, phase II controlled trial. Trials. 2022 Jun 6;23(1):470. doi: 10.1186/s13063-022-06426-2. PMID 35668528
- [Result] Liu J, Lv B, Yin H, Zhu X, Wei H, Ding Y. A Phase I, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose, Multiple Ascending Dose and Food Effect Study to Evaluate the Tolerance, Pharmacokinetics of Jaktinib, a New Selective Janus Kinase Inhibitor in Healthy Chinese Volunteers. Front Pharmacol. 2020 Dec 14;11:604314. doi: 10.3389/fphar.2020.604314. eCollection 2020. PMID 33536914